CLINICAL TRIAL: NCT01443364
Title: Multicenter, Open Label Study to Evaluate the Predictability of Early Response to Certolizumab Pegol (in Combination With Methotrexate) as Confirmed at Week 52 in Subjects With Moderate-severe Rheumatoid Arthritis (RA)
Brief Title: Open Label Study to Assess the Predictability of Early Response to Certolizumab Pegol in Patients With Rheumatoid Arthritis
Acronym: SPEED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Italy s.p.a. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA0069; 2011-000385-35 (EudraCT Number)
Record Dates: First submitted 2011-09-27; First posted 2011-09-29 (Estimated); Results first posted 2016-03-23 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Certolizumab pegol - Cimzia; Rheumatoid Arthritis; Power Doppler Ultrasonography; Italy; Moderate-severe Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Certolizumab pegol (Experimental)
  Interventions: Biological: Certolizumab pegol

INTERVENTIONS:
Biological: Certolizumab pegol — Prefilled syringes containing an injectable volume of 1ml of liquid Certolizumab Pegol (CZP) for single use at a dosage strength of 200 mg/ml. Injections will be given subcutaneously. CZP 400 mg at Week 0, 2 and 4, then continued as maintenance dose of 200 mg every 2 weeks until Week 50.
  Other Names: CIMZIA; CZP

SUMMARY:
The study aims to evaluate the predictability of early response to Certolizumab pegol in combination with Methotrexate at one year in patients with moderate to severe rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of adult-onset Rheumatoid Arthritis (RA) for a duration of at least 6 months but not longer than 5 years
* positive Rheumatoid Factor (RF) and/or positive anti Cyclic Citrullinated Peptide (anti-CCP)
* active RA disease
* subjects must have failed at least one traditional Disease Modifying Anti-Rheumatic Drug (DMARD).
* subject is naïve to RA related biologics

Exclusion Criteria:

* a diagnosis of any other inflammatory arthritis
* history of infected joint prosthesis, or other significant infection
* known Tuberculosis (TB) disease or high risk of acquiring TB infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2011-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (18):
- Italy (18):
  - 11, Bari
  - 08, Catania
  - 10, Ferrara
  - 12, Florence
  - 01, Iesi
  - 05, Milan
  - 13, Milan
  - 18, Milan
  - 07, Modena
  - 23, Monserrato
  - 20, Napoli
  - 16, Padua
  - 06, Roma
  - 21, Roma
  - 22, Siena
  - 09, Torino
  - 04, Udine
  - 02, Verona

REFERENCES:
- [Derived] Sarzi-Puttini P, Filippucci E, Adami S, Meroni PL, Batticciotto A, Idolazzi L, De Lucia O, Talavera P, Kumke T, Grassi W. Clinical, Ultrasound, and Predictability Outcomes Following Certolizumab Pegol Treatment (with Methotrexate) in Patients with Moderate-to-Severe Rheumatoid Arthritis: 52-Week Results from the CZP-SPEED Study. Adv Ther. 2018 Aug;35(8):1153-1168. doi: 10.1007/s12325-018-0751-8. Epub 2018 Jul 24. PMID 30043210
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll patients in December 2011 and concluded in May 2015.
Pre-assignment Details: Participant Flow refers to all subjects randomized who have received at least one dose of study medication.
Groups:
- Certolizumab Pegol: Subjects will be treated for 52 weeks with Certolizumab Pegol (CZP) (administration every two weeks) in combination with Methotrexate (MTX) (administration weekly). Dosing regimen of CZP consists of 3 administrations of 400 mg at Weeks 0, 2 and 4 followed by 200 mg every other week up to and including Week 50.
Period: Overall Study
Arm/Group | Certolizumab Pegol
Started | 132
Completed | 91
Not Completed | 41
Not completed — Lack of Efficacy | 14
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 5
Not completed — Other Reason | 4
Not completed — SAE, non-fatal | 6
Not completed — AE, non-serious non-fatal | 8
Not completed — SAE, non-fatal+AE, non-serious non-fatal | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Characteristics refer to the Safety Set (SS) which consists of all subjects who received at least one dose of study medication.
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 94
  >=65 years | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35
  Not Hispanic or Latino | 97
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kilogram] | 69.33 (14.10)
Height [Mean (Standard Deviation); unit: centimeter] | 164.16 (8.48)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.66 (4.52)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects With Clinical Response at Week 12 Who Also Had Clinical Response at Week 52
Description: Clinical response is defined as a reduction from Baseline (Week 0) of more than 1.2 scores in the Disease Activity Score28 [Erythrocyte Sedimentation Rate] (DAS28-ESR) scoring system
Time Frame: From Baseline to Week 12 and Week 52
Population: The Full Analysis Set (FAS) will consist of all subjects in the Safety Set (SS) who have a valid baseline and valid post-baseline efficacy measurement for the primary variable (DAS28-ESR). One Subject from the SS has been excluded from the FAS Set.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 131
percentage of subjects | 69.1 [58.78 to 78.27]

2. Primary Outcome: The Percentage of Subjects With Clinical Response at Week 8 Who Also Had Clinical Response at Week 52
Description: as for outcome 1
Time Frame: From Baseline to Week 8 and Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 131
percentage of subjects | 69.8 [59.57 to 78.75]

3. Primary Outcome: The Percentage of Subjects With Clinical Response at Week 6 Who Also Had Clinical Response at Week 52
Description: as for outcome 1
Time Frame: From Baseline to Week 6 and Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 131
percentage of subjects | 65.2 [54.33 to 74.96]

4. Primary Outcome: The Percentage of Subjects With Clinical Response at Week 4 Who Also Had Clinical Response at Week 52
Description: as for outcome 1
Time Frame: From Baseline to Week 4 and Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 131
percentage of subjects | 66.7 [56.13 to 76.11]

5. Primary Outcome: The Percentage of Subjects With Clinical Response at Week 2 Who Also Had Clinical Response at Week 52
Description: as for outcome 1
Time Frame: From Baseline to Week 2 and Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 131
percentage of subjects | 64.9 [52.89 to 75.61]

6. Primary Outcome: The Percentage of Subjects With Clinical Response at Week 1 Who Also Had Clinical Response at Week 52
Description: as for outcome 1
Time Frame: From Baseline to Week 1 and Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 131
percentage of subjects | 55.8 [39.88 to 70.92]

7. Secondary Outcome: Change From Baseline in the Synovial Fluid and Proliferation at Week 52
Description: The synovial fluid and proliferation is a semiquantitative score (0-3 on each of 6 joints, with a minimum score of 0 and a maximum score of 18). A greater score indicates greater disease activity.
Time Frame: From Baseline to Week 52
Population: Full Analysis Set (FAS) with Last Observation Carried Forward (LOCF). The FAS will consist of all subjects in the Safety Set who have a valid Baseline and valid post-Baseline efficacy measurement for the primary variable (DAS28-ESR).
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 59
units on a scale | -1.0 [-9 to 4]

8. Secondary Outcome: Change From Baseline in the Synovial Fluid and Proliferation at Week 36
Description: The synovial fluid and proliferation is a semiquantitative score (0-3 on each of 6 joints with a minimum score of 0 and a maximum score of 18). A greater score indicates greater disease activity.
Time Frame: From Baseline to Week 36
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 59
units on a scale | -1.0 [-9 to 4]

9. Secondary Outcome: Change From Baseline in the Synovial Fluid and Proliferation at Week 24
Description: as for outcome 8
Time Frame: From Baseline to Week 24
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 58
units on a scale | -1.0 [-9 to 4]

10. Secondary Outcome: Change From Baseline in the Synovial Fluid and Proliferation at Week 12
Description: as for outcome 8
Time Frame: From Baseline to Week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 58
units on a scale | -1.0 [-12 to 5]

11. Secondary Outcome: Change From Baseline in the Synovial Fluid and Proliferation at Week 8
Description: as for outcome 8
Time Frame: From Baseline to Week 8
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 58
units on a scale | -1.0 [-12 to 2]

12. Secondary Outcome: Change From Baseline in the Synovial Fluid and Proliferation at Week 6
Description: as for outcome 8
Time Frame: From Baseline to Week 6
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 58
units on a scale | -1.0 [-10 to 2]

13. Secondary Outcome: Change From Baseline in the Synovial Fluid and Proliferation at Week 4
Description: as for outcome 8
Time Frame: From Baseline to Week 4
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 58
units on a scale | -1.0 [-8 to 4]

14. Secondary Outcome: Change From Baseline in the Synovial Fluid and Proliferation at Week 2
Description: as for outcome 8
Time Frame: From Baseline to Week 2
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 57
units on a scale | -1.0 [-5 to 4]

15. Secondary Outcome: Change From Baseline in the Synovial Fluid and Proliferation at Week 1
Description: as for outcome 8
Time Frame: From Baseline to Week 1
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 53
units on a scale | 0.0 [-5 to 3]

16. Secondary Outcome: Change From Baseline in the Doppler Signal and Blood Flow at Week 52
Description: The Doppler signal and blood flow is a semiquantitative score (0-3 on each of 6 joints with a minimum score of 0 and a maximum score of 18). A greater score indicates greater disease activity.
Time Frame: From Baseline to Week 52
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 59
units on a scale | -1.0 [-12 to 4]

17. Secondary Outcome: Change From Baseline in the Doppler Signal and Blood Flow at Week 36
Description: as for outcome 16
Time Frame: From Baseline to Week 36
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 59
units on a scale | -1.0 [-11 to 4]

18. Secondary Outcome: Change From Baseline in the Doppler Signal and Blood Flow at Week 24
Description: as for outcome 16
Time Frame: From Baseline to Week 24
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 58
units on a scale | -1.0 [-11 to 6]

19. Secondary Outcome: Change From Baseline in the Doppler Signal and Blood Flow at Week 12
Description: as for outcome 16
Time Frame: From Baseline to Week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 58
units on a scale | -1.0 [-12 to 9]

20. Secondary Outcome: Change From Baseline in the Doppler Signal and Blood Flow at Week 8
Description: as for outcome 16
Time Frame: From Baseline to Week 8
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 58
units on a scale | -1.0 [-12 to 2]

21. Secondary Outcome: Change From Baseline in the Doppler Signal and Blood Flow at Week 6
Description: as for outcome 16
Time Frame: From Baseline to Week 6
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 58
units on a scale | -1.0 [-12 to 2]

22. Secondary Outcome: Change From Baseline in the Doppler Signal and Blood Flow at Week 4
Description: as for outcome 16
Time Frame: From Baseline to Week 4
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 58
units on a scale | -0.5 [-10 to 2]

23. Secondary Outcome: Change From Baseline in the Doppler Signal and Blood Flow at Week 2
Description: as for outcome 16
Time Frame: From Baseline to Week 2
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 57
units on a scale | 0.0 [-10 to 3]

24. Secondary Outcome: Change From Baseline in the Doppler Signal and Blood Flow at Week 1
Description: as for outcome 16
Time Frame: From Baseline to Week 1
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 53
units on a scale | 0.0 [-10 to 3]

25. Secondary Outcome: Change From Baseline in the Cartilage Damage at Week 52
Description: The Cartilage damage is a semiquantitative score (0-4 on each of 6 joints with a minimum score of 0 and a maximum score of 24). A greater score indicates greater disease severity.
Time Frame: From Baseline to Week 52
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 55
units on a scale | 0.0 [-11 to 8]

26. Secondary Outcome: Change From Baseline in the Cartilage Damage at Week 36
Description: as for outcome 25
Time Frame: From Baseline to Week 36
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 55
units on a scale | 0.0 [-12 to 16]

27. Secondary Outcome: Change From Baseline in the Cartilage Damage at Week 24
Description: as for outcome 25
Time Frame: From Baseline to Week 24
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 54
units on a scale | 0.0 [-13 to 11]

28. Secondary Outcome: Change From Baseline in the Cartilage Damage at Week 12
Description: as for outcome 25
Time Frame: From Baseline to Week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 54
units on a scale | 0.0 [-11 to 11]

29. Secondary Outcome: Change From Baseline in the Cartilage Damage at Week 8
Description: as for outcome 25
Time Frame: From Baseline to Week 8
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 54
units on a scale | 0.0 [-11 to 9]

30. Secondary Outcome: Change From Baseline in the Cartilage Damage at Week 6
Description: as for outcome 25
Time Frame: From Baseline to Week 6
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 54
units on a scale | 0.0 [-11 to 7]

31. Secondary Outcome: Change From Baseline in the Cartilage Damage at Week 4
Description: as for outcome 25
Time Frame: From Baseline to Week 4
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 54
units on a scale | 0.0 [-11 to 4]

32. Secondary Outcome: Change From Baseline in the Cartilage Damage at Week 2
Description: as for outcome 25
Time Frame: From Baseline to Week 2
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 53
units on a scale | 0.0 [-11 to 9]

33. Secondary Outcome: Change From Baseline in the Cartilage Damage at Week 1
Description: as for outcome 25
Time Frame: From Baseline to Week 1
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 50
units on a scale | 0.0 [-8 to 4]

34. Secondary Outcome: Change From Baseline in the Bone Erosion at Week 52
Description: The bone erosion is a semiquantitative score (0-4 on each of 6 joints with a minimum score of 0 and a maximum score of 24). A greater score indicates greater disease severity.
Time Frame: From Baseline to Week 52
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 59
units on a scale | 0.0 [-5 to 3]

35. Secondary Outcome: Change From Baseline in the Bone Erosion at Week 36
Description: as for outcome 34
Time Frame: From Baseline to Week 36
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 59
units on a scale | 0.0 [-5 to 4]

36. Secondary Outcome: Change From Baseline in the Bone Erosion at Week 24
Description: as for outcome 34
Time Frame: From Baseline to Week 24
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 58
units on a scale | 0.0 [-5 to 10]

37. Secondary Outcome: Change From Baseline in the Bone Erosion at Week 12
Description: as for outcome 34
Time Frame: From Baseline to Week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 58
units on a scale | 0.0 [-5 to 3]

38. Secondary Outcome: Change From Baseline in the Bone Erosion at Week 8
Description: as for outcome 34
Time Frame: From Baseline to Week 8
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 58
units on a scale | 0.0 [-5 to 5]

39. Secondary Outcome: Change From Baseline in the Bone Erosion at Week 6
Description: as for outcome 34
Time Frame: From Baseline to Week 6
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 58
units on a scale | 0.0 [-5 to 3]

40. Secondary Outcome: Change From Baseline in the Bone Erosion at Week 4
Description: as for outcome 34
Time Frame: From Baseline to Week 4
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 58
units on a scale | 0.0 [-5 to 3]

41. Secondary Outcome: Change From Baseline in the Bone Erosion at Week 2
Description: as for outcome 34
Time Frame: From Baseline to Week 2
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 57
units on a scale | 0.0 [-4 to 2]

42. Secondary Outcome: Change From Baseline in the Bone Erosion at Week 1
Description: as for outcome 34
Time Frame: From Baseline to Week 1
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 53
units on a scale | 0.0 [-4 to 2]

43. Secondary Outcome: Change From Baseline in Sum of the Synovial Fluid and Synovial Proliferation, and Doppler Signal/Blood Flow at Week 52
Description: The sum of the synovial fluid volume, synovial proliferation, Doppler Signal and Blood Flow is a score (0-6 on each of 6 joints with a minimum score of 0 and a maximum score of 36). A greater score indicates greater disease activity.
Time Frame: From Baseline to Week 52
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 59
units on a scale | -3.0 [-20 to 5]

44. Secondary Outcome: Change From Baseline in Sum of the Synovial Fluid and Synovial Proliferation, and Doppler Signal/Blood Flow at Week 36
Description: as for outcome 43
Time Frame: From Baseline to Week 36
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 59
units on a scale | -3.0 [-20 to 6]

45. Secondary Outcome: Change From Baseline in Sum of the Synovial Fluid and Synovial Proliferation, and Doppler Signal/Blood Flow at Week 24
Description: as for outcome 43
Time Frame: From Baseline to Week 24
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 58
units on a scale | -3.0 [-20 to 10]

46. Secondary Outcome: Change From Baseline in Sum of the Synovial Fluid and Synovial Proliferation, and Doppler Signal/Blood Flow at Week 12
Description: as for outcome 43
Time Frame: From Baseline to Week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 58
units on a scale | -3.0 [-23 to 14]

47. Secondary Outcome: Change From Baseline in Sum of the Synovial Fluid and Synovial Proliferation, and Doppler Signal/Blood Flow at Week 8
Description: as for outcome 43
Time Frame: From Baseline to Week 8
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 58
units on a scale | -3.0 [-23 to 3]

48. Secondary Outcome: Change From Baseline in Sum of the Synovial Fluid and Synovial Proliferation, and Doppler Signal/Blood Flow at Week 6
Description: as for outcome 43
Time Frame: From Baseline to Week 6
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 58
units on a scale | -2.5 [-20 to 3]

49. Secondary Outcome: Change From Baseline in Sum of the Synovial Fluid and Synovial Proliferation, and Doppler Signal/Blood Flow at Week 4
Description: as for outcome 43
Time Frame: From Baseline to Week 4
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 58
units on a scale | -2.5 [-17 to 4]

50. Secondary Outcome: Change From Baseline in Sum of the Synovial Fluid and Synovial Proliferation, and Doppler Signal/Blood Flow at Week 2
Description: as for outcome 43
Time Frame: From Baseline to Week 2
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 57
units on a scale | -2.0 [-13 to 4]

51. Secondary Outcome: Change From Baseline in Sum of the Synovial Fluid and Synovial Proliferation, and Doppler Signal/Blood Flow at Week 1
Description: as for outcome 43
Time Frame: From Baseline to Week 1
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 53
units on a scale | -1.0 [-13 to 3]

52. Secondary Outcome: Change From Baseline in the Sum of the Progression in the Doppler Signal, Cartilage Damage and Bone Erosion Score at Week 52
Description: The sum of the progression in the Doppler signal, cartilage damage and bone erosion score is a score (0-11 on each of 6 joints with a minimum score of 0 and a maximum score of 66). A greater score indicates greater disease severity.
Time Frame: From Baseline to Week 52
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 55
units on a scale | -2.0 [-15 to 9]

53. Secondary Outcome: Change From Baseline in the Sum of the Progression in the Doppler Signal, Cartilage Damage and Bone Erosion Score at Week 36
Description: as for outcome 52
Time Frame: From Baseline to Week 36
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 55
units on a scale | -2.0 [-15 to 17]

54. Secondary Outcome: Change From Baseline in the Sum of the Progression in the Doppler Signal, Cartilage Damage and Bone Erosion Score at Week 24
Description: as for outcome 52
Time Frame: From Baseline to Week 24
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 54
units on a scale | -1.5 [-15 to 10]

55. Secondary Outcome: Change From Baseline in the Sum of the Progression in the Doppler Signal, Cartilage Damage and Bone Erosion Score at Week 12
Description: as for outcome 52
Time Frame: From Baseline to Week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 54
units on a scale | -2.0 [-15 to 11]

56. Secondary Outcome: Change From Baseline in the Sum of the Progression in the Doppler Signal, Cartilage Damage and Bone Erosion Score at Week 8
Description: as for outcome 52
Time Frame: From Baseline to Week 8
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 54
units on a scale | -2.0 [-13 to 11]

57. Secondary Outcome: Change From Baseline in the Sum of the Progression in the Doppler Signal, Cartilage Damage and Bone Erosion Score at Week 6
Description: as for outcome 52
Time Frame: From Baseline to Week 6
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 54
units on a scale | -2.0 [-15 to 5]

58. Secondary Outcome: Change From Baseline in the Sum of the Progression in the Doppler Signal, Cartilage Damage and Bone Erosion Score at Week 4
Description: as for outcome 52
Time Frame: From Baseline to Week 4
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 54
units on a scale | -1.0 [-15 to 4]

59. Secondary Outcome: Change From Baseline in the Sum of the Progression in the Doppler Signal, Cartilage Damage and Bone Erosion Score at Week 2
Description: as for outcome 52
Time Frame: From Baseline to Week 2
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 53
units on a scale | -1.0 [-15 to 9]

60. Secondary Outcome: Change From Baseline in the Sum of the Progression in the Doppler Signal, Cartilage Damage and Bone Erosion Score at Week 1
Description: as for outcome 52
Time Frame: From Baseline to Week 1
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 50
units on a scale | -1.0 [-10 to 4]

61. Secondary Outcome: Synovial Fluid and Proliferation at Week 52
Description: as for outcome 8
Time Frame: Week 52
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 65
units on a scale | 5.0 [0 to 16]

62. Secondary Outcome: Synovial Fluid and Proliferation at Week 36
Description: as for outcome 8
Time Frame: Week 36
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 65
units on a scale | 5.0 [0 to 16]

63. Secondary Outcome: Synovial Fluid and Proliferation at Week 24
Description: as for outcome 8
Time Frame: Week 24
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 5.0 [0 to 16]

64. Secondary Outcome: Synovial Fluid and Proliferation at Week 12
Description: as for outcome 8
Time Frame: Week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 5.0 [0 to 13]

65. Secondary Outcome: Synovial Fluid and Proliferation at Week 8
Description: as for outcome 8
Time Frame: Week 8
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 5.0 [0 to 14]

66. Secondary Outcome: Synovial Fluid and Proliferation at Week 6
Description: as for outcome 8
Time Frame: Week 6
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 6.0 [0 to 12]

67. Secondary Outcome: Synovial Fluid and Proliferation at Week 4
Description: as for outcome 8
Time Frame: Week 4
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 6.0 [0 to 13]

68. Secondary Outcome: Synovial Fluid and Proliferation at Week 2
Description: as for outcome 8
Time Frame: Week 2
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 63
units on a scale | 7.0 [0 to 12]

69. Secondary Outcome: Synovial Fluid and Proliferation at Week 1
Description: as for outcome 8
Time Frame: Week 1
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 59
units on a scale | 7.0 [1 to 13]

70. Secondary Outcome: Synovial Fluid and Proliferation at Week 0
Description: as for outcome 8
Time Frame: Week 0 (Baseline)
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 59
units on a scale | 8.0 [0 to 15]

71. Secondary Outcome: Doppler Signal and Blood Flow at Week 52
Description: as for outcome 16
Time Frame: Week 52
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 65
units on a scale | 0.0 [0 to 10]

72. Secondary Outcome: Doppler Signal and Blood Flow at Week 36
Description: as for outcome 16
Time Frame: Week 36
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 65
units on a scale | 0.0 [0 to 10]

73. Secondary Outcome: Doppler Signal and Blood Flow at Week 24
Description: as for outcome 16
Time Frame: Week 24
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 0.0 [0 to 10]

74. Secondary Outcome: Doppler Signal and Blood Flow at Week 12
Description: as for outcome 16
Time Frame: Week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 0.0 [0 to 12]

75. Secondary Outcome: Doppler Signal and Blood Flow at Week 8
Description: as for outcome 16
Time Frame: Week 8
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 0.0 [0 to 7]

76. Secondary Outcome: Doppler Signal and Blood Flow at Week 6
Description: as for outcome 16
Time Frame: Week 6
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 0.5 [0 to 7]

77. Secondary Outcome: Doppler Signal and Blood Flow at Week 4
Description: as for outcome 16
Time Frame: Week 4
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 2.0 [0 to 9]

78. Secondary Outcome: Doppler Signal and Blood Flow at Week 2
Description: as for outcome 16
Time Frame: Week 2
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 63
units on a scale | 1.0 [0 to 11]

79. Secondary Outcome: Doppler Signal and Blood Flow at Week 1
Description: as for outcome 16
Time Frame: Week 1
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 59
units on a scale | 1.0 [0 to 11]

80. Secondary Outcome: Doppler Signal and Blood Flow at Week 0
Description: as for outcome 16
Time Frame: Week 0 (Baseline)
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 59
units on a scale | 2.0 [0 to 12]

81. Secondary Outcome: Cartilage Damage at Week 52
Description: as for outcome 25
Time Frame: Week 52
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 65
units on a scale | 4.0 [0 to 20]

82. Secondary Outcome: Cartilage Damage at Week 36
Description: as for outcome 25
Time Frame: Week 36
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 65
units on a scale | 5.0 [0 to 24]

83. Secondary Outcome: Cartilage Damage at Week 24
Description: as for outcome 25
Time Frame: Week 24
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 4.5 [0 to 19]

84. Secondary Outcome: Cartilage Damage at Week 12
Description: as for outcome 25
Time Frame: Week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 5.0 [0 to 20]

85. Secondary Outcome: Cartilage Damage at Week 8
Description: as for outcome 25
Time Frame: Week 8
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 4.5 [0 to 20]

86. Secondary Outcome: Cartilage Damage at Week 6
Description: as for outcome 25
Time Frame: Week 6
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 63
units on a scale | 4.0 [0 to 20]

87. Secondary Outcome: Cartilage Damage at Week 4
Description: as for outcome 25
Time Frame: Week 4
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 63
units on a scale | 4.0 [0 to 20]

88. Secondary Outcome: Cartilage Damage at Week 2
Description: as for outcome 25
Time Frame: Week 2
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 61
units on a scale | 4.0 [0 to 21]

89. Secondary Outcome: Cartilage Damage at Week 1
Description: as for outcome 25
Time Frame: Week 1
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 57
units on a scale | 5.0 [0 to 21]

90. Secondary Outcome: Cartilage Damage at Week 0
Description: as for outcome 25
Time Frame: Week 0 (Baseline)
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 56
units on a scale | 6.0 [0 to 21]

91. Secondary Outcome: Bone Erosion at Week 52
Description: as for outcome 34
Time Frame: Week 52
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 65
units on a scale | 2.0 [0 to 10]

92. Secondary Outcome: Bone Erosion at Week 36
Description: as for outcome 34
Time Frame: Week 36
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 65
units on a scale | 2.0 [0 to 11]

93. Secondary Outcome: Bone Erosion at Week 24
Description: as for outcome 34
Time Frame: Week 24
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 2.0 [0 to 11]

94. Secondary Outcome: Bone Erosion at Week 12
Description: as for outcome 34
Time Frame: Week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 2.0 [0 to 10]

95. Secondary Outcome: Bone Erosion at Week 8
Description: as for outcome 34
Time Frame: Week 8
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 2.0 [0 to 10]

96. Secondary Outcome: Bone Erosion at Week 6
Description: as for outcome 34
Time Frame: Week 6
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 2.0 [0 to 10]

97. Secondary Outcome: Bone Erosion at Week 4
Description: as for outcome 34
Time Frame: Week 4
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 2.0 [0 to 10]

98. Secondary Outcome: Bone Erosion at Week 2
Description: as for outcome 34
Time Frame: Week 2
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 63
units on a scale | 2.0 [0 to 15]

99. Secondary Outcome: Bone Erosion at Week 1
Description: as for outcome 34
Time Frame: Week 1
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 59
units on a scale | 2.0 [0 to 15]

100. Secondary Outcome: Bone Erosion at Week 0
Description: as for outcome 34
Time Frame: Week 0 (Baseline)
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 60
units on a scale | 2.0 [0 to 15]

101. Secondary Outcome: Sum of the Synovial Fluid and Synovial Proliferation, and Doppler Signal/Blood Flow at Week 52
Description: as for outcome 43
Time Frame: Week 52
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 65
units on a scale | 5.0 [0 to 26]

102. Secondary Outcome: Sum of the Synovial Fluid and Synovial Proliferation, and Doppler Signal/Blood Flow at Week 36
Description: as for outcome 43
Time Frame: Week 36
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 65
units on a scale | 6.0 [0 to 26]

103. Secondary Outcome: Sum of the Synovial Fluid and Synovial Proliferation, and Doppler Signal/Blood Flow at Week 24
Description: as for outcome 43
Time Frame: Week 24
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 6.5 [0 to 26]

104. Secondary Outcome: Sum of the Synovial Fluid and Synovial Proliferation, and Doppler Signal/Blood Flow at Week 12
Description: as for outcome 43
Time Frame: Week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 7.0 [0 to 22]

105. Secondary Outcome: Sum of the Synovial Fluid and Synovial Proliferation, and Doppler Signal/Blood Flow at Week 8
Description: as for outcome 43
Time Frame: Week 8
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 6.0 [0 to 16]

106. Secondary Outcome: Sum of the Synovial Fluid and Synovial Proliferation, and Doppler Signal/Blood Flow at Week 6
Description: as for outcome 43
Time Frame: Week 6
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 7.0 [0 to 16]

107. Secondary Outcome: Sum of the Synovial Fluid and Synovial Proliferation, and Doppler Signal/Blood Flow at Week 4
Description: as for outcome 43
Time Frame: Week 4
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 8.0 [0 to 18]

108. Secondary Outcome: Sum of the Synovial Fluid and Synovial Proliferation, and Doppler Signal/Blood Flow at Week 2
Description: as for outcome 43
Time Frame: Week 2
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 63
units on a scale | 8.0 [0 to 23]

109. Secondary Outcome: Sum of the Synovial Fluid and Synovial Proliferation, and Doppler Signal/Blood Flow at Week 1
Description: as for outcome 43
Time Frame: Week 1
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 59
units on a scale | 8.0 [1 to 23]

110. Secondary Outcome: Sum of the Synovial Fluid and Synovial Proliferation, and Doppler Signal/Blood Flow at Week 0
Description: as for outcome 43
Time Frame: Week 0 (Baseline)
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 59
units on a scale | 10.0 [1 to 24]

111. Secondary Outcome: Sum of the Progression in the Doppler Signal, Cartilage Damage and Bone Erosion Score at Week 52
Description: as for outcome 52
Time Frame: Week 52
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 65
units on a scale | 7.0 [0 to 38]

112. Secondary Outcome: Sum of the Progression in the Doppler Signal, Cartilage Damage and Bone Erosion Score at Week 36
Description: as for outcome 52
Time Frame: Week 36
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 65
units on a scale | 8.0 [0 to 38]

113. Secondary Outcome: Sum of the Progression in the Doppler Signal, Cartilage Damage and Bone Erosion Score at Week 24
Description: as for outcome 52
Time Frame: Week 24
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 10.0 [0 to 38]

114. Secondary Outcome: Sum of the Progression in the Doppler Signal, Cartilage Damage and Bone Erosion Score at Week 12
Description: as for outcome 52
Time Frame: Week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 9.0 [0 to 38]

115. Secondary Outcome: Sum of the Progression in the Doppler Signal, Cartilage Damage and Bone Erosion Score at Week 8
Description: as for outcome 52
Time Frame: Week 8
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 64
units on a scale | 9.0 [0 to 34]

116. Secondary Outcome: Sum of the Progression in the Doppler Signal, Cartilage Damage and Bone Erosion Score at Week 6
Description: as for outcome 52
Time Frame: Week 6
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 63
units on a scale | 8.0 [0 to 33]

117. Secondary Outcome: Sum of the Progression in the Doppler Signal, Cartilage Damage and Bone Erosion Score at Week 4
Description: as for outcome 52
Time Frame: Week 4
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 63
units on a scale | 8.0 [0 to 34]

118. Secondary Outcome: Sum of the Progression in the Doppler Signal, Cartilage Damage and Bone Erosion Score at Week 2
Description: as for outcome 52
Time Frame: Week 2
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 61
units on a scale | 10.0 [0 to 43]

119. Secondary Outcome: Sum of the Progression in the Doppler Signal, Cartilage Damage and Bone Erosion Score at Week 1
Description: as for outcome 52
Time Frame: Week 1
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 57
units on a scale | 10.0 [0 to 47]

120. Secondary Outcome: Sum of the Progression in the Doppler Signal, Cartilage Damage and Bone Erosion Score at Week 0
Description: as for outcome 52
Time Frame: Week 0 (Baseline)
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 55
units on a scale | 12.0 [0 to 47]

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events were reported from Baseline (Week 0) up to the Safety Follow-up Visit (Week 60).
Description: Adverse Events refer to the Safety Set (SS) which consists of all subjects who received at least one dose of study medication.
Arm/Group | Certolizumab Pegol
Serious Adverse Events (participants affected / at risk) | 16/132
Other Adverse Events (participants affected / at risk) | 31/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (N=132)
Retroperitoneal lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Periorbital oedema (Eye disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Endophthalmitis (Infections and infestations) | 1 (1)
Paratyphoid fever (Infections and infestations) | 1 (1)
Lobular breast carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anosmia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Bladder mass (Renal and urinary disorders) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Genital prolapse (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (N=132)
Pyrexia (General disorders) | 7 (7)
Influenza (Infections and infestations) | 15 (16)
Bronchitis (Infections and infestations) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days